CLINICAL TRIAL: NCT02076321
Title: The Effect of NSAID Use in the Acute Phase of Skeletally Immature Bone Healing: A Prospective Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Daniel Hoernschemeyer, Orthopaedic Surgeon, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1207111
Record Dates: First submitted 2014-02-19; First posted 2014-03-03 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-01

CONDITIONS: Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Acetaminophen; Ibuprofen

ARMS (2):
- Acetaminophen (Other): control group
  Interventions: Drug: Acetaminophen
- NSAID (Ibuprofen) (Other): Study group
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — acetaminophen for pain control with dose and frequency of 10-15mg/kg/dose, Maximum dose 1000mg. Maximum amount per day: 75mg/kg (not to exceed 4g/day).
  Other Names: Tylenol
  Arms: Acetaminophen
Drug: Ibuprofen — ibuprofen for pain control with dose and frequency 4-10mg/kg/dose. Maximum of 40mg/kg/day, not to exceed 3,200mg/day. Maximum one-time dose of 800mg.
  Other Names: Advil; Motrin
  Arms: NSAID (Ibuprofen)

SUMMARY:
Non-steroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen, are excellent medications for providing pain control in children with fractures or those who have surgery to correct bony deformity requiring the bone to be cut (osteotomy) and realigned. There is some data to suggest that these types of medications can adversely affect bone healing in adult patients with broken bones or those having spine fusion surgery. There is little data with regard to how these medications effect bone healing in children. With this project, the investigators' goal is to determine if NSAIDs delay or otherwise adversely effect bone healing and to demonstrate that these medications adequately control pain in children with broken bones or those who have had an osteotomy.

DETAILED DESCRIPTION:
Non-steroidal anti-inflammatory drugs (NSAIDs) are effective in controlling both post-operative pain and pain associated with orthopaedic injuries, particularly in the pediatric population. Additionally, use of NSAIDs for pain control in this setting avoids the use of narcotic pain medications, the adverse effects of which are well known.

Recent research has suggested a possible association between use of NSAIDs and impaired fracture healing in the skeletally mature, or adult, population. Several adult mammal studies have demonstrated inhibition of bony repair with administration of NSAIDs. Yet, other adult animal studies have failed to find the same effect. Clinical data in the adult population is similarly conflicted, with some studies showing an inhibition of bone healing after posterior spinal fusion, while a larger study found no correlation. The data investigating the effects of NSAID use in adults after fracture or osteotomy is even less clear with some studies demonstrating higher rates of non-union with NSAID administration and others finding no significant effect on bone healing.

The research investigating these outcomes in the skeletally immature population is limited; one study compared administration of ketorolac versus normal saline for 7, 14 and 21 days in a juvenile rat model with a stabilized tibia fracture. They found no significant difference in strength, stiffness or histological characteristics of fracture callus between the two groups. Clinical retrospective studies of the pediatric population with regard to use of NSAIDs after posterior spinal fusion have failed to reproduce findings of inhibitory effects on bone healing. Similarly, two retrospective studies found no cases of delayed union or non-union in pediatric patients who received perioperative ketorolac around the time of operative fixation of fractures, or osteotomy. Given these results, the way in which and the degree to which NSAIDs perturb the inflammatory mileu during the acute phase of healing is potentially distinct from the effects on bone healing in the skeletally mature.

There have been no clinical prospective, randomized studies to evaluate the effect, if any, that NSAIDs have on bone healing in the skeletally immature patient population. The investigators hypothesize that NSAID administration in the acute phase of bone healing, whether it be a fracture or osteotomy, will not result in delayed union or non-union as compared to patients who take acetaminophen for pain control during this same time period.

ELIGIBILITY:
Inclusion Criteria:

* • Male aged 16 years or less or female aged 14 years or less

  * Open physis on radiographs
  * Fracture undergoing closed treatment or operative treatment or patient undergoing elective osteotomy

Exclusion Criteria:

* • Regular use of NSAIDs

  * Allergy to NSAIDs
  * Inability to take breakthrough medications due side effects or allergy
  * Systemic illness
  * Renal impairment
  * Liver disease
  * Polytrauma
  * Uncontrolled diabetes
  * Regular use of corticosteroids
  * History of any skeletal dysplasia
  * History of neuromuscular disorder
  * History of bleeding disorder
  * History of liver disorder
  * Pathologic fracture
  * Closed physes
  * Male greater than 16 years old
  * Female greater than 14 years old
  * Pregnant or possibly pregnant females based on report and last menstrual period

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Hoernschemeyer, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health System, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetaminophen | NSAID (Ibuprofen)
Started | 51 | 51
Completed | 46 | 49
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | NSAID (Ibuprofen) | Total
Number analyzed (Participants) | 46 | 49 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 49 | 95
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 7.44 [2 to 16] | 7.67 [1.5 to 16] | 7.56 [1.5 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Compare the Time to Union of Fractures and Osteotomies in Skeletally Immature Patients Administered NSAIDs for Pain Control, Versus Those Administered Acetaminophen for Pain Control.
Time Frame: The subject will be enrolled/assessed up to 6 months post-injury/osteotomy.
Measure: Mean (Full Range); unit: Days
Arm/Group | Acetaminophen | NSAID (Ibuprofen)
Number analyzed (Participants) | 51 | 51
Days | 41.2 [22 to 84] | 40.5 [19 to 98]

ADVERSE EVENTS:
Arm/Group | Acetaminophen | NSAID (Ibuprofen)
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes